CLINICAL TRIAL: NCT06269887
Title: Dominant and Non-Dominant Upper Extremity in Young Individuals
Brief Title: Dominant Non-Dominant Upper Extremity in Gender
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Study director, PT, PhD, Karabuk University
Other Study IDs: Karabuk-001
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Upper Extremity Problem; Gender Issues
MeSH Terms: conditions — Sexism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male: Hand preference was evaluated with the Edinburgh Hand Preference Questionnaire, grip muscle strength with the Jamar dynamometer, dexterity with the Purdue Pegboard Test, and proprioception as joint position sense with the inclinometer.
- Female: Hand preference was evaluated with the Edinburgh Hand Preference Questionnaire, grip muscle strength with the Jamar dynamometer, dexterity with the Purdue Pegboard Test, and proprioception as joint position sense with the inclinometer.

SUMMARY:
There are strength and functional differences between non-dominant and dominant extremities. This is important in the hand and extremity rehabilitation process. This situation also differs between genders. Comparison of the dominant and non-dominant limb can provide important clinical or rehabilitation field-related information. It is reported in the literature that manual dexterity, grip strength and joint position sense may differ between extremities. However, the relationship between this situation and the difference between genders has not been explained. It is thought that examining this difference can be extremely useful in determining achievable goals in hand rehabilitation and in customizing care for different groups.

DETAILED DESCRIPTION:
Many treatment protocols compare the strength of the injured extremity to the uninjured extremity or compare it to normative data from the same group of individuals. There is controversy about the difference in grip strength between dominant and non-dominant hands in left- and right-hand dominant individuals. There is no study in the literature that evaluates the differences in muscle strength, joint position sense and upper extremity function skills between dominant and non-dominant upper extremities between genders. It is very important to include bilateral activity training in rehabilitation programs that aim to improve upper extremity mobility and speed. In addition, it will contribute to the accurate evaluation of activity and participation limitations, the determination of priorities, the selection of the right activity in task-specific and target-oriented treatment approaches, and the achievement of more effective results when integrated with technology-supported approaches. Therefore, the aim of our study is to fill this gap in the literature by comparing the differences between dominant and non-dominant upper extremities between genders.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-25
2. Volunteering to participate in the study

Exclusion Criteria:

1. Having trauma (fracture, dislocation) in the last year
2. Doing sports or activities that require bilateral activity (playing music, knitting, sports, etc.)
3. Being diagnosed with any neurological or orthopedic disease that will affect hand-eye coordination
4. Having had upper extremity surgery
5. Having any Botox injection in the last 6 months
6. Those who did not agree to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adult individuals will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Hand Preference | First Day
  The Edinburgh Hand Preference Questionnaire questions individuals' hand use in daily living activities. The final total score is between 100 and -100. Individuals who score more than 40 points are right-hand; Individuals in this score range from 40 to -40 inclusive are recorded as ambidextrous, and individuals with scores of -40 points and below are left-handed
Grip Strength | First Day
  Hand grip strength was measured using a standard Jamar Dynamometer.
Joint Position Sense | First Day
  Proprioception was assessed by joint position sense (JPS) test. Shoulder JPS was assessed using a digital inclinometer
Manual Dexterity | First Day
  The Purdue Pegboard Test was used to evaluate the functional skill levels of the upper extremities.

CONTACTS AND LOCATIONS:
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhat AK, Jindal R, Acharya AM. The influence of ethnic differences based on upper limb anthropometry on grip and pinch strength. J Clin Orthop Trauma. 2021 Jul 15;21:101504. doi: 10.1016/j.jcot.2021.101504. eCollection 2021 Oct. PMID 34367910
- [Result] Amo-Setien FJ, Leal-Costa C, Abajas-Bustillo R, Gonzalez-Lamuno D, Redondo-Figuero C; EXERNET Research Group. Factors associated with grip strength among adolescents: An observational study. J Hand Ther. 2020 Jan-Mar;33(1):96-102. doi: 10.1016/j.jht.2018.10.005. Epub 2018 Nov 30. PMID 30503041
- [Result] Dag F, Erdogan AT. Gender and age differences in absolute and relative handgrip strength of the Turkish population aged 8-27 years. Hand Surg Rehabil. 2020 Dec;39(6):556-563. doi: 10.1016/j.hansur.2020.06.005. Epub 2020 Aug 18. PMID 32818689